CLINICAL TRIAL: NCT04322617
Title: Anlotinib With or Without Immune Checkpoint Inhibitors in Standard Chemo-immunotherapy Failed Advanced Non-small Cell Lung Cancer
Brief Title: Anlotinib Plus Immune Checkpoint Inhibitors for Lung Cancer
Acronym: ATHENA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200113
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Anlotinib, Immune Checkpoint Inhibitor, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: Anlotinib with the same Immune Checkpoint Inhibitors. (Experimental): Anlotinib plus Immune Checkpoint Inhibitors which has been used in first line treatment.
  Interventions: Drug: Anlotinib plus the same Immune Checkpoint Inhibitors.
- Cohort B: Anlotinib with the new Immune Checkpoint Inhibitors. (Experimental): Anlotinib plus Immune Checkpoint Inhibitors which has not been used in first line treatment.
  Interventions: Drug: Anlotinib plus the new Immune Checkpoint Inhibitors.
- Cohort C: Anlotinib Monotherapy. (Experimental): Anlotinib Monotherapy.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib plus the same Immune Checkpoint Inhibitors. — Anlotinib, 8mg po qd, D1-D14 every 21days.
  Other Names: Pembrolizumab, Sintilimab etc. have been used in the previous treatment.
  Arms: Cohort A: Anlotinib with the same Immune Checkpoint Inhibitors.
Drug: Anlotinib plus the new Immune Checkpoint Inhibitors. — Anlotinib, 8mg po qd, D1-D14 every 21days.
  Other Names: Pembrolizumab, Sintilimab etc. have not been used in the previous treatment.
  Arms: Cohort B: Anlotinib with the new Immune Checkpoint Inhibitors.
Drug: Anlotinib — Anlotinib, 8mg po qd, D1-D14 every 21days.
  Other Names: Anlotinib monotherapy.
  Arms: Cohort C: Anlotinib Monotherapy.

SUMMARY:
This study aims to explore the efficacy of Anlotinib with or without Immune Checkpoint Inhibitor in Standard Chemo-immunotherapy Failed Advanced NSCLC.

DETAILED DESCRIPTION:
This study aims to explore the efficacy of Anlotinib with or without Immune Checkpoint Inhibitor in Standard Chemo-immunotherapy Failed Advanced NSCLC. The primary endpoint was PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histopathology or cytology confirmed lung cancer
4. Failed from first line Chemo-immunotherapy.
5. ECOG 0-1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.
9. Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

1. Subjects who have received any of the following treatments must be excluded:

   * Treatment with molecules such as EGFR, VEGFR antibodies within 4 weeks prior to the first dose of study drug.
   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
   * Ongoing (or inability to discontinue) possibly potent CYP1A2, CYP3A inhibitor (1 week), or inducer (2 weeks) drug therapy or herbal supplements within 1-2 weeks prior to the first dose.
2. Presence of spinal cord compression or meningeal metastasis.
3. History of other malignant tumors within 2 years.
4. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
5. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
6. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
7. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
8. Heart-related diseases or abnormalities
9. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
10. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
11. Live vaccine was given 2 weeks before the first medication.
12. Women who are breastfeeding or pregnant.
13. Hypersensitivity to the test drug and the ingredients.
14. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2028-03-24 (Estimated); Study Completion 2029-03-24 (Estimated)

PRIMARY OUTCOMES:
Progression free survival time (PFS) | Time from first subject dose to study completion, or up to 36 month.
  Progression free survival time define as first dose to first documented disease progression assessed by investigator or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 month.
  Objective response rate define as the proportion of subjects who have a complete response (CR) or a partial response (PR).
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month.
  To assess overall survival, define as first dose to the death of the subject due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China